CLINICAL TRIAL: NCT06130943
Title: Evaluation of the Quality of Telephone Calls to a Suicide Prevention Helpline
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B6702020000210
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Suicide Prevention; Suicidal Ideation
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study adds to the existing evidence on suicide prevention helpline efficacy because it tackles some of the common limitations for helpline studies. High risk individuals were not excluded from the study, since there was no human interference in deciding if the study was offered to the lifeline callers. Most of the existing studies exclude users in high risk and acute crisis situations. The study employed the callers' own ratings on a set of questions, automatically offered within the phone system immediately before and after the call to assess the immediate impact of the call and the intervention. The automatization of the self-report measures in the telephone system reduces the burden on the operators to offer the research questions without interrupting the crisis intervention and decreases the risk of bias in caller responses.

The goal of this observational study is to evaluatie the Flesmish suicide prevention helpline in people who call the helpline when feeling suicidal. The main questions it aims to answer are:

1. Has the degree to which the caller feels in crisis subsided? (Crisis in this is seen as the subjective feeling of complete emotional upset)
2. Does the caller report feeling less suicidal? (Score on selected indicators of suicidality, particularly hopelessness, entrapment, controllability, suicidal intent and social support)
3. Is the caller satisfied with the conversation?
4. Which elements in the conversation (i.e., responders' interventions) make it more or less effective, in terms of crisis level, suicidality (indicators) and caller satisfaction?
5. Which elements of the conversation do callers name as (not) helpful during the follow-up conversation? Which elements promoted progress in this, besides merely lowering the crisis level?
6. What possible (follow-up) actions do callers see as helping to sustain and/or improve the longer-term impact of the conversation with the suicide prevention helpline?

Participants are asked the fill in items before the call, immediately after the call and one to two weeks after the call.

DETAILED DESCRIPTION:
All adult (18+) callers who contact the suicide prevention helpline are offered the opportunity to participate in the study, once per (coded) phone number. The study is presented to the caller before there is any interaction between the caller and the operator and only when an operator is immediately available to answer the call. Informed consent is acquired in two steps, in order to minimise the time between calling and being transferred to the operator for callers not wanting to participate in the study: callers are asked if they are interested in taking part in the research: if not, they are transferred immediately to the operator; if they indicated being interested they receive more information about the study. The information about the study, which is recorded, is given automatically by the telephone system. Callers can consent by using the telephone keypad. More detailed information about the study is available for them on the website of the helpline.

After consenting, participants are asked about their age and gender and to respond to six short statements on their state of crisis and suicidality. All questions are answered using the telephone keys. After completing the questionnaire, or whenever they want to discontinue the study, participants are immediately transferred to the operator.

At the end of the call, a post-test is offered to the participants using the automatic telephone system. The six statements on the state of crisis and suicidality are assessed again, in addition a question on the degree of satisfaction with the call. After completing the post-test participants are asked whether they want to participate in the follow-up study. In order to contact them a phone number on which they can be contacted after one to two weeks, is asked. This phone number is coded by the phone system in order to guarantee the anonymity of the participant.

One to two weeks after contacting the helpline, a follow-up interview is conducted. This interview is carried out by an interviewer with extensive training in crisis calls. After making an initial contact with the participant, the six statements on the state of crisis and suicidality and the satisfaction about the call are assessed again automatically.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years of age or older
* Dutch-speaking
* calling to the Flemish suicide prevention helpline because they felt suicidal

Only callers for whom it is certain that they will be connected to the Flemish suicide prevention helpline will be asked to participate.

Exclusion Criteria:

* Third party callers were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All callers who contact the suicide prevention helpline are asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 608 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Indicatorts of crisis and suicidality | Baseline, post (immediately after the call), follow-up (one to two weeks after the call)
  Since there is no common standardized set of measures for suicide prevention helplines (Mazzer et al., 2021; Trail et al., 2022) six indicators of suicidal ideation and behaviour (SIB) are used to evaluate the calls of the Flemish Suicide Prevention Helpline. The selection of the indicators is based on previous research on helpline efficacy (Gould et al., 2007; Hoffberg et al., 2020; Hvidt et al., 2016; Kalafat et al., 2007), and on a number of core elements identified in suicide prevention theories explaining the transition from suicidal ideation to suicidal behaviour. The six indicators are crisis, hopelessness, entrapment, controllability, suicidal intent, and social support. All indicators are scored by the callers on a 10-point Likert scale (using the telephone keypad), ranging from 0 (not at all) to 9 (totally).

SECONDARY OUTCOMES:
Satisfaction with the service | Post (immediately after the call), follow-up (one to two weeks after the call)
  The satisfaction of the caller is assessed by the question 'I am satisfied about the call I just had with the suicide prevention helpline'.

OTHER OUTCOMES:
Follow-up interview | Follow-up (one to two weeks after the call)
  Semi-structured interview assessing quality and effectiveness of, and satisfaction with, the conversation at the suicide prevention helpline

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Suicide Prevention, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided